CLINICAL TRIAL: NCT06833372
Title: Extracorporeal Shock Wave Therapy in Patients With Knee Arthritis
Brief Title: Shock Waves in Knee Arthritis
Acronym: SWinKA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SWinKA
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Arthritis of Knee
Keywords: shock waves; conservative treatment
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Prospective randomized clinical study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Active Comparator): only a daily exercise program for 4 weeks: passive and active assisted movement of the knee joint, hamstring stretching, and quadriceps strengthening exercises
  Interventions: Other: exercise group
- ESWT group (Experimental): Shockwave therapy will be administered using an ESWT device (Minilith SL1, Storz) once a week for three consecutive weeks, for a total of three sessions. A focused shockwave modality with an electromagnetic device was chosen for the therapy.
  Interventions: Device: ESWT group

INTERVENTIONS:
Device: ESWT group — During each session, participants will receive 2000 pulses at a frequency of 4 Hz and an EDF between 0.02 and 0.2 mJ/mm2.
  Other Names: shock waves therapy
  Arms: ESWT group
Other: exercise group — daily exercise program
  Other Names: exercise
  Arms: Exercise Group

SUMMARY:
Pathological arthritis is a degenerative disease affecting the joints, characterized by pain, limitation of movement up to ankylosis and disability. Treatment is aimed at reducing pain and slowing the loss of functionality of the district. Among conservative treatments, pharmacological options (NSAIDs, cortisone, contrasupplements, hyaluronic acid) and non-pharmacological options (therapeutic exercise, physical therapy, orthosis, etc.) are indicated. In cases not responding to conservative treatments, surgical treatment will be necessary with prosthetic replacement of the joint district.

DETAILED DESCRIPTION:
In recent years, shock wave therapy has received a lot of interest in the treatment of numerous musculoskeletal pathologies. This physical therapy exploits the cavitational effect induced on the tissues which translates into neo-angiogenic, anti-inflammatory, regenerative and analgesic action. Until now, the indication has been reserved for the treatment of tendinopathies and delayed consolidation of fractures. Pre-clinical research is also paving the way for the treatment of cartilage pathologies; in fact, after the stimulation of the chondrocyte, a modulation of the phlogogenic cytokines has been found, supporting a slowing down of the progression of the arthritic pathology. The first clinical experiences on arthritic models, such as rhizarthrosis, allow to support the indication also on the pathological model of gonarthrosis. The aim of this study is to verify the effects of shock wave therapy in the patient affected by gonarthrosis, monitoring the action on pain, functionality and tissue district changes.

ELIGIBILITY:
Inclusion Criteria:

* persistent knee pain for at least 3 months, measured with a VAS scale of 4 or higher,
* clinical and radiological diagnosis confirming knee osteoarthritis grade 2 and 3 based on the Kellgren-Lawrence system,
* no history of physical therapy in the last 3 months,
* no infections, tumors in the treatment area of the knee,
* no pathology other than osteoarthritis that could cause knee pain,
* no pathology of the lumbar spine or hip that could refer knee pain,
* free from any condition that prevents participation in exercise or physical therapy willing to participate regularly in the treatment programs were included in the study.

Exclusion Criteria:

* inability to walk,
* a history of clinically symptomatic spinal stenosis or lumbar radiculopathy,
* evidence of a neurological disorder based on history or physical examination,
* generalized pain or fibromyalgia,
* secondary osteoarthritis (to metabolic or rheumatologic disease),
* administration of intra-articular injections (anesthetic, hyaluronic acid, cortisone) of the knee in the last 6 months,
* use of NSAIDs, paracetamol or topical agents in the previous week,
* a previous history of surgery involving the knee joint,
* contraindications to physical therapy (PM, epilepsy, neoplasia, coagulopathy, pregnancy).

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
recovery of pain | From enrollment to 1, 3 and 6 months
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | From enrollment to 1, 3 and 6 months
  questionnaire consisting of 24 questions addressing pain, stiffness and physical function. Score from 0 to 96, higher scores correspond to worse clinical condition.

SECONDARY OUTCOMES:
Roles and Maudsley Score | At 1, 3 and 6 months
  rating of the perception of one's own clinical improvement, from 1 (excellent) to 4 (poor).
MR image | From enrollment to 6 months
  weighted in t2 according to the ICRS classification

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico di Bari, Bari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao Z, Ji H, Jing R, Liu C, Wang M, Zhai L, Bai X, Xing G. Extracorporeal shock-wave therapy reduces progression of knee osteoarthritis in rabbits by reducing nitric oxide level and chondrocyte apoptosis. Arch Orthop Trauma Surg. 2012 Nov;132(11):1547-53. doi: 10.1007/s00402-012-1586-4. Epub 2012 Jul 24. PMID 22825641
- [Background] Ochiai N, Ohtori S, Sasho T, Nakagawa K, Takahashi K, Takahashi N, Murata R, Takahashi K, Moriya H, Wada Y, Saisu T. Extracorporeal shock wave therapy improves motor dysfunction and pain originating from knee osteoarthritis in rats. Osteoarthritis Cartilage. 2007 Sep;15(9):1093-6. doi: 10.1016/j.joca.2007.03.011. Epub 2007 Apr 26. PMID 17466542
- [Background] Mostafa MSEM, Hamada HA, Kadry AM, Zahran SS, Helmy NA. Effect of High-Power Laser Therapy Versus Shock Wave Therapy on Pain and Function in Knee Osteoarthritis Patients: A Randomized Controlled Trial. Photobiomodul Photomed Laser Surg. 2022 Mar;40(3):198-204. doi: 10.1089/photob.2021.0136. Epub 2022 Jan 5. PMID 34986012